CLINICAL TRIAL: NCT00041717
Title: Double-Blind, Placebo-Controlled, 12-Week Parallel Group Study to Evaluate Safety and Efficacy of Oral Fampridine-SR in Subjects With Moderate to Severe Spasticity Resulting From Chronic, Incomplete Spinal Cord Injury
Brief Title: Safety and Efficacy of Oral Fampridine-SR for the Treatment of Spasticity Resulting From Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCI-F301
Record Dates: First submitted 2002-07-12; First posted 2002-07-16 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2013-04

CONDITIONS: Spinal Cord Injury; Muscle Spasticity
Keywords: spinal cord injury; muscle spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fampridine-SR 50mg/day (Active Comparator)
  Interventions: Drug: Fampridine-SR
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fampridine-SR — 25mg bid (twice daily)
  Arms: fampridine-SR 50mg/day
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with spinal cord injury, some fibers may be destroyed at the site of injury, while others remain connected but do not work correctly to carry electrical impulses. As a result, subjects with an incomplete spinal cord injury may have spasticity which is muscle spasms or muscle stiffness that makes movement difficult. Fampridine-SR is an experimental drug that increases the ability of the nerve to conduct electrical impulses. This study will examine the effects of Fampridine-SR on moderate to severe lower-limb spasticity, as well as the effects on bodily functions such as bladder control, bowel function and sexual function. The study will also examine the possible risks of taking Fampridine-SR.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete traumatic Spinal Cord Injury (at least 18 months prior and stable for 6 months)
* Moderate to severe lower-limb spasticity
* Able to give informed consent and willing to comply with protocol

Exclusion Criteria:

* Pregnancy
* History of seizures
* Existing or history of frequent Urinary Tract Infections
* History of drug or alcohol abuse
* Allergy to pyridine-containing substances
* Received a botox injection 4 months prior to study
* Received an investigational drug within 30 days
* Previously treated with 4-aminopyridine (4-AP)
* Not on stable medication dosing in 3 weeks prior to study
* Abnormal ECG or laboratory value at screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2002-07; Primary Completion 2004-02 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blight, Study Director — Acorda Therapeutics
Locations (45):
- United States (37):
  - Lakeshore Rehabilitation Hospital, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Baptist Medical Center, Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, California
  - Neuro-Therapeutics, Inc, Pasadena, California
  - Neurology Associates, P.A., Wilmington, Delaware
  - National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Miami Center to Cure Paralysis at the Univ. of Miami School of Medicine, Miami, Florida
  - Rehabilitation Hospital, Sunrise, Florida
  - Shepherd Spinal Center, Atlanta, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center-Dept. of Physical Medicine & Rehabilitation-EMG, Oak Lawn, Illinois
  - Springfield Clinic-Neuroscience Institute, Springfield, Illinois
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - HEALTHSOUTH Braintree Rehabilitation Hospital, Braintree, Massachusetts
  - HEALTHSOUTH New England Rehabilitation Hospital, Woburn, Massachusetts
  - Mary Free Bed Hospital & Rehabilitation Center, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, Div. of Rehab/Neurology, St Louis, Missouri
  - Montana Neuroscience, Missoula, Montana
  - Kessler Institute of Rehabilitation, West Orange, New Jersey
  - The Burke Rehabilitation Hospital, White Plains, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Clinical Research Services, Bismarck, North Dakota
  - Drake Center, Cincinnati, Ohio
  - Cleveland VAMC, Cleveland, Ohio
  - Good Shepherd Rehabilitation, Allentown, Pennsylvania
  - Bryn Mawr Rehabilitation Hospital, Malvern, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - HEALTHSOUTH Harmarville Rehabilitation Hospital, Pittsburgh, Pennsylvania
  - Northeastern Rehabilitation Associates, Scranton, Pennsylvania
  - Rehabilitation Services University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Hampton VA Hospital, Hampton, Virginia
  - Richmond VA Medical Center (Hunter Holmes McGuire), Richmond, Virginia
  - CAMC Health Education & Research Institute, Charleston, West Virginia
- Canada (8):
  - Foothills Provincial General Hospital, Calgary, Alberta
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - G.F. Strong Rehabilitation Centre, Vancouver, British Columbia
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - QEII HSC-Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia
  - Parkwood Hospital Site, St. Joseph's Health Care, London, Ontario
  - The Rehabilitation Centre, Ottawa, Ontario
  - Toronto Rehabilitation Institute, Lyndhurst Centre, Toronto, Ontario

REFERENCES:
- See also: Related Info — http://www.acorda.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population consists of patients with chronic incomplete spinal cord injury (SCI) whose injury occurred at least 18 months prior to screening, and whose neurological status has been stable for at least 6 months.
Pre-assignment Details: One patient did not take any investigational drug and was excluded from the safety and ITT populations. The remaining 212 patients were included in the ITT and safety populations: 98 in the placebo and 114 in the Fampridine-SR 25 mg b.i.d. group.
Groups:
- Fampridine-SR 50mg/Day: Fampridine-sustained release (SR) : 25mg bid (twice daily)
- Placebo: Placebo : Placebo
Period: Overall Study
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Started | 114 | 98
Completed | 81 | 86
Not Completed | 33 | 12

BASELINE CHARACTERISTICS:
Groups:
- Fampridine-SR 50mg/Day: Fampridine-SR : 25mg bid (twice daily)
- Total: Total of all reporting groups
Arm/Group | Fampridine-SR 50mg/Day | Placebo | Total
Number analyzed (Participants) | 114 | 98 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.05) | 40.1 (13.10) | 40.9 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 100 | 85 | 185
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 12 | 30
  White | 94 | 81 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Change From Baseline in Ashworth Score Evaluating Spasticity
Description: The Ashworth Score is the average rating (based on a scale of 1 to 5) of four lower extremity muscle groups; left and right knee flexors and extensors (hamstrings and quadriceps muscles). A higher Ashworth Score indicates a greater degree of abnormal muscle tone (spasticity) and a negative change in score indicates improvement.
Time Frame: Baseline (visits 2,3) average score days 7,14 and double blind treatment period (visits 4-7) average score days 28-98
Population: Intent to treat (ITT) population
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 109 | 96
units on a scale | -0.19 (0.039) | -0.15 (0.042)

2. Primary Outcome: Double-blind Change From Baseline in Subject's Global Impression (SGI) of Treatment
Description: This questionnaire asked the patient to evaluate the effects of investigational drug on his/her quality of life during the preceding week using a 7-point scale (from 1=terrible to 7=delighted). A positive change score in SGI indicates improved outcome.
Time Frame: Baseline (visits 2,3) average score days 7,14 and double blind treatment period (visits 4-7) average score days 28-98
Population: ITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Number analyzed (Participants) | 109 | 96
units on a scale | -0.2 (0.08) | -0.1 (0.09)

ADVERSE EVENTS:
Time Frame: Treatment-emergent serious adverse events (SAE) include SAEs with date of onset (or worsening) on or after the start of double-blind treatment and no more than 30 days after the last dose of investigational drug.
Arm/Group | Fampridine-SR 50mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 6/114 | 6/98
Other Adverse Events (participants affected / at risk) | 94/114 | 84/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR 50mg/Day (N=114) | Placebo (N=98)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Reaction unevaluable (General disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertonia (Psychiatric disorders) | 0 (0) | 1 (1)
Hyperesthesia (Psychiatric disorders) | 1 (2) | 0 (0)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary incontinence (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR 50mg/Day (N=114) | Placebo (N=98)
Urinary tract infection (Infections and infestations) | 34 (42) | 16 (20)
Hypertonia (Nervous system disorders) | 23 (31) | 25 (35)
Constipation (Gastrointestinal disorders) | 11 (18) | 8 (9)
Dizziness (Vascular disorders) | 15 (18) | 3 (4)
Pain (General disorders) | 13 (18) | 14 (18)
Accidental injury (Injury, poisoning and procedural complications) | 10 (17) | 17 (19)
Headache (Nervous system disorders) | 10 (15) | 8 (13)
Dyspepsia (Gastrointestinal disorders) | 8 (12) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (12) | 4 (5)
Asthenia (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (6)
Infection (Infections and infestations) | 9 (11) | 10 (12)
Paresthesia (Nervous system disorders) | 10 (11) | 5 (5)
Sweating (Skin and subcutaneous tissue disorders) | 7 (11) | 1 (1)
Insomnia (Psychiatric disorders) | 10 (10) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 (10) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 8 (8)
Nervousness (Psychiatric disorders) | 8 (8) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (12)
Pelvic pain (Renal and urinary disorders) | 5 (7) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 3 (7) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 1 (1)
Chills (General disorders) | 4 (6) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 6 (6) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Depression (Psychiatric disorders) | 5 (5) | 4 (4)
Fever (General disorders) | 5 (5) | 2 (2)
Hypotonia (Nervous system disorders) | 4 (5) | 1 (1)
Confusion (Psychiatric disorders) | 3 (4) | 0 (0)
Flu syndrome (Infections and infestations) | 4 (4) | 4 (4)
Gastroenteritis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 2 (2)
Abnormal gait (General disorders) | 3 (3) | 1 (1)
Amblyopia (Eye disorders) | 3 (3) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3) | 2 (3)
Hyperesthesia (Nervous system disorders) | 2 (3) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Peripheral edema (General disorders) | 3 (3) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (4)
Chest pain (General disorders) | 1 (1) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 3 (5)
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 6 (6)
Vesiculobullous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.